CLINICAL TRIAL: NCT07005310
Title: Ultra Long Peripheral Catheter Versus Accelerated Seldinger Technique Long Peripheral Catheter in Difficult Intravenous Access Patients: a Pragmatic Randomised Controlled Trial
Brief Title: Ultra-Long Peripheral Catheter Versus Accelerated Seldinger Technique Long Peripheral Catheter in Difficult IV Access Patients
Acronym: ULAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, Tim Torsy, Prof. Dr., University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2024-0303
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Difficult Intravenous Access; Adults
Keywords: Long peripheral catheter; Accelerated seldinger technique; Pragmatic randomized controlled trial; Dwell time; complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated seldinger technique LPC (Active Comparator): One study arm will be assigned the AST-long peripheral catheter (Powerglide Pro long peripheral catheter, BD) available in 18G 100 mm, 20G 100 mm (approx. 3.94 inches) and 22G 80 mm (approx. 3.15 inches).
  Interventions: Device: Powerglide pro™
- Ultra-long peripheral catheter (Experimental): The other study arm will be assigned the ultralong peripheral catheter (Introcan Safety deep access catheter, B. Braun) available in 18, 20 and 22G and 63.5 mm (approx. 2.5 inches) in length.
  Interventions: Device: Introcan safety deep access

INTERVENTIONS:
Device: Powerglide pro™ — A long peripheral catheter will be placed under ultrasound guidance. This catheter will be placed by using the Accelerated seldinger technique.
  Arms: Accelerated seldinger technique LPC
Device: Introcan safety deep access — The catheter will be placed using ultrasound guidance and by using the 'catheter-over-the needle' approach.
  Arms: Ultra-long peripheral catheter

SUMMARY:
The aim of this study is to perform a comparative analysis of clinical outcomes associated with the use of an ultra-long peripheral catheter using (catheter-over-the-needle technique) versus an AST-long peripheral catheter in adult patients with difficult intravenous access (DIVA) in a real-world clinical setting. Specifically, the study will assess potential benefits, including longer mean catheter dwell time and improved catheter usability, as well as potential harms, such as increased incidence of catheter-related thrombosis, infections, phlebitis, infiltration, and unplanned catheter removal.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients with DIVA, requiring placement of a long peripheral catheter, will be included in the study.
* A digital request form for venous access must be completed by the treating physician at the ward.
* Patients must be proficient in either Dutch or French
* Patients must have decision-making capacity or be represented by a legal representative.

Exclusion Criteria:

* Expected therapy duration of less than 24 hours
* pregnancy
* Need for central venous access
* Inability to locate a deep peripheral vein in the upper extremity prior enrollment in the study
* Veins located deeper than 1.6cm prior enrollment in the study
* withdrawal of consent, or presentation at a time when study personnel are unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dwell time | Until study completion, an average of 14 days.
  is defined as the duration between the date of catheter insertion and the date of its removal, expressed in hours.

SECONDARY OUTCOMES:
Number of Participants with Catheter related thrombosis | Until study completion, an average of 14 days.
  CRT indicates the presence of clots in the vascular system after the placement of a catheter due to induced trauma to the endothelium, inflammation, individual patient factors and catheter related factors. The following types of thrombi will be reported.
  * Mural thrombus or Obstructive thrombus
  * Symptomatic or asymptomatic thrombus
Number of Participants with Midline catheter related infections | Until study completion, an average of 14 days.
  MLABSI are defined as laboratory confirmed bloodstream infections in patients who had a midline catheter in place for two or more calendar days prior to confirmation. MLABSI will be diagnosed as:
  * differential time to positivity >2 h in comparing cultures blood samples drawn from the catheter and from a peripheral vein if the catheter is fully patent
  * isolation of the same microorganism (species and antimicrobial susceptibility testing) from the catheter tip (>15 colony forming units) and a peripheral blood sample if blood draws are impossible
  These parameters will be combined to report MLABSI.
Number of Participants with Phlebitis | Until study completion, an average of 14 days.
  Phlebitis will be defined as the inflammation of a vein resulting from mechanical, chemical, or bacterial causes. The severity of this inflammation will be assessed using the Visual Infusion Phlebitis (VIP) scale, which assigns a score ranging from 0 to 5, with 0 indicating a healthy insertion site. A score of 5 on the VIP scale signifies severe pain, redness, palpable venous cord, and fever-related complaints. A score of 2, indicating pain, erythema and swelling, necessitates immediate catheter relocation. Symptomatic catheter-related thrombosis must be excluded in advance.
Number of Participants with Loss of catheter usability | Until study completion, an average of 14 days.
  Loss of catheter usability will be registered by using the following categories38:
  Total occlusion: inability to infuse and aspirate Sub-occlusion: Difficulty in infusing and aspirating Persistent withdrawal occlusion: No blood withdrawal possibility
Number of Participants with Unplanned removal | Until study completion, an average of 14 days.
  Removal of an uncomplicated catheter without therapy completion (accidental removal, patient death)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
The data is confidential.

REFERENCES:
- [Derived] Pieteraerens W, Vanhonacker D, Beeckman K, Torsy T. Ultra long peripheral catheter versus accelerated Seldinger technique long peripheral catheter in difficult intravenous access patients (ULAST): a pragmatic randomised controlled trial protocol. BMJ Open. 2026 Feb 6;16(2):e106079. doi: 10.1136/bmjopen-2025-106079. PMID 41651529